CLINICAL TRIAL: NCT02661347
Title: Transcranial Direct Current Stimulation for Hallucinations in First-Episode Schizophrenia
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty in recruiting patients who met the eligibility criteria.
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, Deepak Sarpal, Psychiatrist, Northwell Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB# 15-0701
Record Dates: First submitted 2016-01-20; First posted 2016-01-22 (Estimated); Last update posted 2018-03-13 (Actual); Status verified 2018-03

CONDITIONS: Schizophrenia; Schizophreniform; Schizoaffective Disorder; Psychosis Not Otherwise Specified (NOS)
Keywords: First Episode; Schizophreniform; Schizoaffective Disorder; Psychosis; Schizophrenia; tDCS; Risperidone; Anti-psychotic medication
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Risperidone; Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active comparator: tDCS & Risperidone (Active Comparator): In the active arm, active tDCS will be applied using a Soterix Medical 1x1 line tDCS Model 1300 low-intensity stimulator at a current of 2 milliampere (mA) for 20 minutes, twice a day for five consecutive days, for a total of 10 sessions.
  Interventions: Drug: Risperidone; Device: tDCS
- Sham comparator: tDCS & Risperidone (Sham Comparator): In the sham arm, active tDCS will be applied using a Soterix Medical 1x1 line tDCS Model 1300 low-intensity stimulator at a current of 2mA for 1 minute, twice a day for five consecutive days, for a total of 10 sessions.
  Interventions: Drug: Risperidone; Device: tDCS

INTERVENTIONS:
Drug: Risperidone — The dosage for risperidone will be 1 mg to 6 mg per day. The dose of the risperidone will be based on the participant's clinical improvement and side effects.
Device: tDCS — Transcranial direct current stimulation (tDCS) is a form of non-invasive brain stimulation in which sub-threshold transcranial electric current (in the range of 0.4-2 mA) is applied via two conductive saline soaked electrodes placed on the scalp using a Soterix Medical 1x1 line tDCS Model 1300 low-intensity stimulator.

SUMMARY:
The purpose of this study is to test the efficacy of transcranial direct current stimulation (tDCS) for the treatment of auditory hallucinations in patients currently on risperidone treatment who are experiencing recent onset psychosis.

DETAILED DESCRIPTION:
This study looks to investigate whether patients with recent onset psychosis may benefit from tDCS treatment. The main hypothesis to be tested in this study is that treatment with risperidone supplemented with tDCS will yield a decrease in auditory hallucinations and negative symptoms; and improve working memory and attention.

To test this hypothesis the investigators will enroll 30 patients with recent-onset psychosis into a 16-week long randomized double blind controlled study of risperidone treatment supplemented with tDCS versus risperidone plus sham tDCS. Patients who present for treatment of a first psychotic episode with a schizophrenia spectrum diagnosis and who are eligible to undergo or are already on treatment with risperidone, will be randomized to either tDCS or sham tDCS twice a day for five consecutive days. Neuropsychological testing, Magnetic Resonance Imaging (MRI) and electroencephalogram (EEG) will be conducted at baseline, week 1 (after completion of tDCS or sham tDCS intervention) and week 16. Clinical interviews to assess symptoms and medical assessments for side effects will be done at baseline, weekly for the first four weeks and then every two weeks until study completion. The primary outcome measure will be the Auditory Hallucinations Rating Scale (AHRS) score.

Specific aims are:

To determine the efficacy of tDCS for auditory hallucinations in patients with first episode schizophrenia. The investigators hypothesize that risperidone plus tDCS is associated with a faster and more robust decrease in auditory hallucinations compared to risperidone plus sham tDCS.

To test the efficacy of tDCS in cognitive and negative symptoms in patients with first episode schizophrenia. The investigators hypothesize that tDCS improves working memory, attention/vigilance and decreases negative symptoms.

To examine the neuronal basis of tDCS effects in ameliorating auditory hallucinations in schizophrenia by conducting event-related potential (ERP) and resting state EEG. The investigators hypothesize that the Delta N-100 amplitude is associated with improvement of auditory hallucinations after tDCS treatment.

To determine the effects of tDCS on brain structure and function by conducting structural MRI, diffusion tensor imaging (DTI) and functional magnetic resonance imaging (fMRI).

ELIGIBILITY:
Inclusion Criteria:

1. current Diagnostic and Statistical Manual-IV (DSM-IV) -defined diagnosis of schizophrenia, schizophreniform, schizoaffective disorder, psychosis NOS as assessed using the Structured Clinical Interview for Axis I DSM-IV Disorders (SCID-I/P) (First et al, 1994).
2. does not meet DSM-IV criteria for a current substance-induced psychotic disorder, a psychotic disorder due to a general medical condition, delusional disorder, brief psychotic disorder, shared psychotic disorder, or a mood disorder with psychotic features.
3. current positive symptoms rated ≥4 (moderate) on one or more of these BPRS (Woerner et al., 1988) items: conceptual disorganization, grandiosity, hallucinatory behavior, unusual thought content
4. current positive symptoms rated ≥4 (moderate) on one or more of these BPRS (Woerner et al., 1988) items: conceptual disorganization, grandiosity or unusual thought content and is in the first episode of the illness as defined by having taken antipsychotic medications for a cumulative lifetime period of 4 weeks or less,
5. age 15 to 40.
6. competent and willing to sign informed consent.
7. for women, negative pregnancy test and agreement to use a medically accepted birth control method.

Exclusion Criteria:

1. serious neurological or endocrine disorder or any medical condition or treatment known to affect the brain.
2. any medical condition which requires treatment with a medication with psychotropic effects.
3. significant risk of suicidal or homicidal behavior;
4. cognitive or language limitations, or any other factor that would preclude subjects providing informed consent.
5. medical contraindications to treatment with risperidone (e.g. neuroleptic malignant syndrome with prior risperidone exposure).
6. lack of response to a prior adequate trial of risperidone.
7. requires treatment with an antidepressant or mood stabilizing medication.
8. presence of an electrically, magnetically or mechanically activated implant (including cardiac pacemaker), an intracerebral vascular clip, or any other electrically sensitive support system.
9. damaged skin at the site of stimulation (i.e. skin with ingrown hairs, acne, razor nicks, wounds that have not healed, recent scar tissue, broken skin, etc.).

Ages: 15 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2016-02; Primary Completion 2016-12-01 (Actual); Study Completion 2016-12-01 (Actual)

PRIMARY OUTCOMES:
Auditory hallucinations | 16 Weeks
  A decrease in verbal auditory hallucinations based on the Auditory Hallucinations Ratings Scale (AHRS).

CONTACTS AND LOCATIONS:
Overall Officials: Deepak Sarpal, M.D., Principal Investigator — Northwell Health
Locations (1):
- Zucker-Hillside Hospital, Glen Oaks, New York, United States

IPD SHARING:
Plan to Share IPD: No